CLINICAL TRIAL: NCT03406117
Title: A Study to Determine the Dermatological Safety and Sensitizing Potential of HAT1 Topical Products Using Cumulative Irritation, Phototoxicity, and Repeated Insult Patch Tests
Brief Title: A Study to Determine the Safety and Sensitizing Potential of HAT1 Topical Products Using Skin Sensitivity Patch Tests
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haus Bioceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HCTP16MD0204
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Healthy; Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- HAT1-EPBF2 (Experimental): CIT was conducted over a period of approximately 15 days for each subject to determine the irritation and/or sensitization potential of a test material(s) under occlusion by 14 repeated closed occlusive patch application every 24 hrs. A final grade was taken 24 hours following the last patch application.
  PT was conducted over a period of approximately 6 days for each subject to determine the phototoxicity of the test product.
  HRIPT was conducted over a period of approximately 6-8 weeks for each subject to confirm that the test substances will not produce evidence of delayed contact sensitization following external contact with the skin by means of a repeated patch application procedure.
  Interventions: Drug: HAT1
- HAT1-HMF3 (Experimental): CIT was conducted over a period of approximately 15 days for each subject to determine the irritation and/or sensitization potential of a test material(s) under occlusion by 14 repeated closed occlusive patch application every 24 hrs. A final grade was taken 24 hours following the last patch application.
  PT was conducted over a period of approximately 6 days for each subject to determine the phototoxicity of the test product.
  HRIPT was conducted over a period of approximately 6-8 weeks for each subject to confirm that the test substances will not produce evidence of delayed contact sensitization following external contact with the skin by means of a repeated patch application procedure.
  Interventions: Drug: HAT1
- Saline Solution: Sodium Chloride (Active Comparator): Saline, Sodium Chlorine (NaCl; 0.9%), was used as the negative irritant control in the CIT portion of the study
  Interventions: Other: Saline Solution

INTERVENTIONS:
Drug: HAT1 — All the participants will have the test product applied to the appropriate test sites by trained study staff. The study was conducted on a mixed population comprising of normal subjects, and patients with atopic dermatitis and active plaque psoriasis.
  Other Names: HAT01
  Arms: HAT1-EPBF2; HAT1-HMF3
Other: Saline Solution — Only for CIT portion of the study. Participant will have product applied topically on site by the trained study staff.
  Other Names: Sodium Chloride
  Arms: Saline Solution: Sodium Chloride

SUMMARY:
The objective of this clinical study is to assess the irritation and sensitisation potential of HAT1 topical products after repeated patch applications to healthy human participants by following conventional Repeated Insult (HRIPT), Cumulative Irritation (CIT), and Phototoxicity (PT) methodologies under the supervision of dermatologists.

DETAILED DESCRIPTION:
For HRIPT, a total of 9 induction patches were applied at the rate of three patches per week for three weeks. The patch was retained in place for 48 hours during week days and 72 hrs over the weekend. Each induction patch was applied to the same site unless the degree of reaction to the test substance or the adhesive necessitates relocation. Two sites, adjacent to the original site, were available if patch relocation was deemed necessary. A rest period of 12-20 days between the final induction patch application and challenge patch application was provided. Challenge patches were applied 12-20 days after the last induction patch application. Patches were worn for 48 hours (± 1 hour), then removed at the site and discarded.

For PT, the test products along with a blank chamber as negative control were applied on the back of the subjects in contralateral paired symmetry under occlusion for 24 hours. After completion of 24 hours of occlusion, both patch systems were taken off. Subjects were acclimatized for 30 minutes post removal of the patch and dermatological assessment of the sites (including controls) was performed. Post assessment, one of the two sites and an untreated blank control site (randomized and investigator blinded) was irradiated with 0.5 MED (specific for each subject). Follow up assessments were performed at 10 minutes post irradiation and subsequently at 24 and 48 hours post irradiation.

For CIT, the patches were prepared in a vertical row and applications were made every day for 14 days. All applications for individual test substances were made to the same site (the site used for the initial patch application) unless reactions become so strong (grade of 2.0 or greater) as to make continued application inadvisable. Patches were worn for approximately 23 hours (± 1 hour). Subjects were instructed to keep their patches dry. Subjects were instructed to return to the test facility for patch removal and disposal by test facility personnel. Skin sites were gently wiped with water and patted dry to remove excess test substance immediately following patch removal. Skin sites were graded approximately 20-40 minutes following patch removal. Subjects were not allowed to replace any patches that fall off. Subjects were provided with instructions and a schedule of the study dates on the first day of the study. Telephone numbers were provided to report adverse events or answer questions on a 24-hour basis.

ELIGIBILITY:
The study population in this report comprises of healthy normal subjects, patients with active plaque psoriasis, and patients with atopic dermatitis.

Inclusion Criteria:

* Males or females 18 years of age or older - no more than 20% of the panel should be comprised of subjects over the age of 65.
* In general good health as determined by the Medical and Dermatological History Questionnaire, or as having diagnosed with atopic dermatitis confirmed by the investigating dermatologist, or as having diagnosed with active plaque psoriasis confirmed by the investigating dermatologist.
* Able to read, understand and sign an informed consent agreement after being advised of the nature of the study.
* Willing to refrain from using lotions, creams, powders or other skin preparations on the skin in the test area for the duration of the study.
* Willing to refrain from exposing skin sites to the sun or going to tanning beds for the duration of the study.

Exclusion Criteria:

* Have a clinical diagnosis of a dermatological condition other that atopic dermatitis or psoriasis (such as contact dermatitis, cutaneous lymphoma, tinea corpori's, etc.), or have non plaque forms of psoriasis (for example, erythrodermic, guttate, or pustular), or have bacterial infections of the skin, including impetigo or abscesses.
* Have a history of skin cancer or have received treatment (chemotherapy, radiation, immune suppressant medications) for any type of cancer within the last 6 months.
* Have a condition or are taking medication(s) which, in the judgment of the Investigator or Designate, makes the subject ineligible or places the subject at undue risk.
* Have pigmentation, extensive scarring, or pigmented lesions in the patch areas, which could interfere with the scoring.
* Have had a mastectomy or axillary lymph nodes removed.
* Have an autoimmune or immune deficiency disease (e.g. lupus, myositis, Crohns disease, autoimmune thyroid diseases, autoimmune hepatitis, etc.).
* Are currently taking any immunosuppressant medication 8. Have insulin-dependent diabetes.
* Have asthma or any other chronic respiratory condition requiring daily therapy
* Are currently using on a routine or frequent basis antihistamines or any systemic or topical anti-inflammatory medications (e.g. ibuprofen, corticosteroid, etc.). Maximum acceptable dosage should be determined by written laboratory guidelines.
* Have used a topical anti-inflammatory in the patch area within the last 2 weeks
* Are currently receiving allergy injections, expects to start injections before the conclusion of the study or has had the final injection within a week of the study start
* Are currently participating in another dermal study of any kind
* Are currently participating in any clinical study, which in the judgment of the Investigator or Designate, could potentially affect responses in either study.
* Have a confirmed skin allergy as a result of participation in a patch study.
* Have a known sensitivity or allergy relating to the substance(s) being evaluated.
* Have a known sensitivity or allergy to adhesives, surgical tapes, bandages, etc.
* Have scars, moles, sunburn, tattoos, etc. in the patch area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-06-26 (Actual); Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
Visual assessment (Patch assessment) | Upto Week 8
  An overall average skin grade is calculated (i.e. the sum of the daily average skin grades divided by the number of study days) for each test substance. An overall skin grade is a representation of average skin reaction during the study.

CONTACTS AND LOCATIONS:
Overall Officials: P Alex, M.D., Study Director — Study Director